CLINICAL TRIAL: NCT01634100
Title: A Randomised, Open-label, Three-way Crossover Trial to Investigate the Effect of Rifampicin and Probenecid on Empagliflozin Pharmacokinetics in Healthy Male and Female Subjects
Brief Title: Drug-interaction Trial in Healthy Subjects With Oral Administration of Empagliflozin (BI 10773), Rifampicin and Probenecid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1245.83; 2012-000971-17 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — Probenecid; Rifampin; empagliflozin

ARMS (3):
- A (Reference) (Experimental): Empagliflozin (BI 10773), Film-coated tablet, single dose
  Interventions: Drug: Probenecid; Drug: Empagliflozin; Drug: Rifampicin
- B (Test 1) (Experimental): Empagliflozin (BI 10773), Film-coated tablet, single dose, and Rifampicin,Film-coated tablet single dose
  Interventions: Drug: Rifampicin; Drug: Empagliflozin
- C (Test 2) (Experimental): Empagliflozin (BI 10773), Film-coated tablet, single dose, and Probenecid Tablet twice daily
  Interventions: Drug: Probenecid; Drug: Empagliflozin (BI 10773)

INTERVENTIONS:
Drug: Probenecid — Probenecid
  Arms: A (Reference)
Drug: Rifampicin — Rifampicin
  Arms: B (Test 1)
Drug: Empagliflozin — BI Drug
  Arms: A (Reference)
Drug: Empagliflozin — BI Drug
  Arms: B (Test 1)
Drug: Rifampicin — Rifampicin
  Arms: A (Reference)
Drug: Probenecid — Probenecid
  Arms: C (Test 2)
Drug: Empagliflozin (BI 10773) — BI Drug
  Arms: C (Test 2)

SUMMARY:
The objectives of the trial are to investigate the effect of concurrent administration of rifampicin and probenecid on the pharmacokinetics of empagliflozin.

ELIGIBILITY:
Inclusion criteria:

1. healthy male and female subjects

Exclusion criteria:

1. any relevant deviation from healthy conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.83.1 Boehringer Ingelheim Investigational Site, Biberach, Germany

REFERENCES:
- [Derived] Macha S, Koenen R, Sennewald R, Schone K, Hummel N, Riedmaier S, Woerle HJ, Salsali A, Broedl UC. Effect of gemfibrozil, rifampicin, or probenecid on the pharmacokinetics of the SGLT2 inhibitor empagliflozin in healthy volunteers. Clin Ther. 2014 Feb 1;36(2):280-90.e1. doi: 10.1016/j.clinthera.2014.01.003. Epub 2014 Feb 1. PMID 24491572

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a randomised, 3-way crossover trial. 18 patients were randomised to one of six treatment sequences and treated. It was an open label trial in which each treatment period lasted 4 days with a washout period of at least 7 days between each.
Groups:
- Empa Alone / Empa + Rifampicin / Empa + Probenecid: Patients were administered three treatments in the following order:
  * Empa Alone (A single dose of 10mg of empagliflozin (empa))
  * Empa + Rifampicin (A single dose of 10mg empagliflozin (empa) combined with a single dose of 600 mg rifampicin)
  * Empa + Probenecid (A single dose of 10mg empagliflozin (empa) in the morning of day 1 combined with 500 mg of probenecid given twice daily for four days from day -1 to day 3)
- Empa Alone / Empa + Probenecid / Empa + Rifampicin: Patients were administered three treatments in the following order:
  * Empa Alone (A single dose of 10mg of empagliflozin (empa))
  * Empa + Probenecid (A single dose of 10mg empagliflozin (empa) in the morning of day 1 combined with 500 mg of probenecid given twice daily for four days from day -1 to day 3)
  * Empa + Rifampicin (A single dose of 10mg empagliflozin (empa) combined with a single dose of 600 mg rifampicin)
- Empa + Rifampicin / Empa Alone / Empa + Probenecid: Patients were administered three treatments in the following order:
  * Empa + Rifampicin (A single dose of 10mg empagliflozin (empa) combined with a single dose of 600 mg rifampicin)
  * Empa Alone (A single dose of 10mg of empagliflozin (empa))
  * Empa + Probenecid (A single dose of 10mg empagliflozin (empa) in the morning of day 1 combined with 500 mg of probenecid given twice daily for four days from day -1 to day 3)
- Empa + Rifampicin / Empa + Probenecid / Empa Alone: Patients were administered three treatments in the following order:
  * Empa + Rifampicin (A single dose of 10mg empagliflozin (empa) combined with a single dose of 600 mg rifampicin)
  * Empa + Probenecid (A single dose of 10mg empagliflozin (empa) in the morning of day 1 combined with 500 mg of probenecid given twice daily for four days from day -1 to day 3)
  * Empa Alone (A single dose of 10mg of empagliflozin (empa))
- Empa + Probenecid / Empa Alone / Empa + Rifampicin: Patients were administered three treatments in the following order:
  * Empa + Probenecid (A single dose of 10mg empagliflozin (empa) in the morning of day 1 combined with 500 mg of probenecid given twice daily for four days from day -1 to day 3)
  * Empa Alone (A single dose of 10mg of empagliflozin (empa))
  * Empa + Rifampicin (A single dose of 10mg empagliflozin (empa) combined with a single dose of 600 mg rifampicin)
- Empa + Probenecid / Empa + Rifampicin / Empa Alone: Patients were administered three treatments in the following order:
  * Empa + Probenecid (A single dose of 10mg empagliflozin (empa) in the morning of day 1 combined with 500 mg of probenecid given twice daily for four days from day -1 to day 3)
  * Empa + Rifampicin (A single dose of 10mg empagliflozin (empa) combined with a single dose of 600 mg rifampicin)
  * Empa Alone (A single dose of 10mg of empagliflozin (empa))
Period: Overall Study
Arm/Group | Empa Alone / Empa + Rifampicin / Empa + Probenecid | Empa Alone / Empa + Probenecid / Empa + Rifampicin | Empa + Rifampicin / Empa Alone / Empa + Probenecid | Empa + Rifampicin / Empa + Probenecid / Empa Alone | Empa + Probenecid / Empa Alone / Empa + Rifampicin | Empa + Probenecid / Empa + Rifampicin / Empa Alone
Started | 3 | 3 | 3 | 3 | 3 | 3
Received Empa Alone | 3 | 3 | 3 | 3 | 3 | 3
Received Empa + Rifampicin | 3 | 3 | 3 | 3 | 3 | 3
Received Empa + Probenecid | 2 | 3 | 2 | 3 | 3 | 3
Completed | 2 | 3 | 2 | 3 | 3 | 3
Not Completed | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set. Total number of patients randomised and treated in the study.
Groups:
- Study Overall: This was a randomised, 3-way crossover trial. 18 patients were randomised to one of six treatment sequences and treated. It was an open label trial in which each treatment period lasted 4 days with a washout period of at least 7 days between each.
Arm/Group | Study Overall
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Total Empagliflozin: Area Under the Curve 0 to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of total empagliflozin (empa) in plasma over the time interval from 0 extrapolated to infinity.
Time Frame: 15 minutes (min) prior to the first dose and 20min, 40min, 1 hour (h), 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h and 72h after the first dose
Population: Pharmacokinetic (PK) set: The PK analysis set includes all subjects who took at least 1 dose of investigational treatment and provided at least 1 evaluable observation for at least 1 primary PK endpoint in at least 1 treatment period without any important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Groups:
- Empa Alone: A single dose of 10mg of empagliflozin (empa).
- Empa + Rifampicin: A single dose of 10mg empagliflozin (empa) combined with a single dose of 600 mg rifampicin.
- Empa + Probenecid: A single dose of 10mg empagliflozin (empa) in the morning of day 1 combined with 500 mg of probenecid given twice daily for four days from day -1 to day 3.
Arm/Group | Empa Alone | Empa + Rifampicin | Empa + Probenecid
Number analyzed (Participants) | 18 | 18 | 16
nmol*h/L | 2240 (28.1) | 3020 (28.2) | 3400 (28.7)
Statistical Analysis 1: Comparison: Empa Alone vs Empa + Rifampicin; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa and rifampicin divided by empa; ANOVA; Based on an ANOVA including the random effect subjects within sequences and the fixed effects sequence, period and treatment; Geometric Mean Ratio = 135.20, 90% CI 2-sided [129.58 to 141.06], Standard Deviation 7.3 — Standard deviation is actually the intra-subject coefficient of variation
Statistical Analysis 2: Comparison: Empa Alone vs Empa + Probenecid; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus probenecid divided by empa; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 153.47, 90% CI 2-sided [146.41 to 160.88], Standard Deviation 7.4 — Standard deviation is actually the intra-subject coefficient of variation

2. Primary Outcome: Total Empa: Maximum Measured Concentration (Cmax)
Description: Maximum measured concentration of total empa in plasma, per period.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Empa Alone | Empa + Rifampicin | Empa + Probenecid
Number analyzed (Participants) | 18 | 18 | 16
nmol/L | 301 (31.6) | 527 (27.5) | 373 (30.9)
Statistical Analysis 1: Comparison: Empa Alone vs Empa + Rifampicin; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa and rifampicin divided by empa; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 175.14, 90% CI 2-sided [160.14 to 191.56], Standard Deviation 15.4 — Standard deviation is actually the intra-subject coefficient of variation
Statistical Analysis 2: Comparison: Empa Alone vs Empa + Probenecid; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus probenecid divided by empa; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 125.60, 90% CI 2-sided [113.67 to 138.78], Standard Deviation 15.9 — Standard deviation is actually the intra-subject coefficient of variation

3. Secondary Outcome: Total Empagliflozin: Area Under the Curve 0 to Time of Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of total empagliflozin (empa) in plasma over the time interval from 0 extrapolated to the time of last the quantifiable data point.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Empa Alone | Empa + Rifampicin | Empa + Probenecid
Number analyzed (Participants) | 18 | 18 | 16
nmol*h/L | 2200 (28.6) | 3000 (28.4) | 3350 (29.1)
Statistical Analysis 1: Comparison: Empa Alone vs Empa + Rifampicin; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa and rifampicin divided by empa; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 136.42, 90% CI 2-sided [130.61 to 142.48], Standard Deviation 7.5 — Standard deviation is actually the intra-subject coefficient of variation
Statistical Analysis 2: Comparison: Empa Alone vs Empa + Probenecid; Test type: Non-Inferiority or Equivalence — Ratio calculated as empa plus probenecid divided by empa; ANOVA; [statistical method as in outcome 1, analysis 1]; Geometric Mean Ratio = 153.61, 90% CI 2-sided [146.50 to 161.06], Standard Deviation 7.5 — Standard deviation is actually the intra-subject coefficient of variation

ADVERSE EVENTS:
Time Frame: Treatment period until end of washout period/end of study examination, up to 29 days
Arm/Group | Empa Alone | Empa + Rifampicin | Empa + Probenecid
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 7/18 | 9/18 | 6/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empa Alone (N=18) | Empa + Rifampicin (N=18) | Empa + Probenecid (N=16)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 2
Vomiting (Gastrointestinal disorders) | 2 | 3 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 3 | 5 | 3
Presyncope (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.